CLINICAL TRIAL: NCT02276794
Title: The Effects of Thrust Versus Non-thrust Manipulation on Pain, Trunk Proprioception and Postural Stability in Subjects With Chronic Low Back Pain
Brief Title: Thrust Versus Non-thrust Manipulation in Chronic Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Time and funding constraints
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Giovanni Esteves Ferreira, PT, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19051513.5.0000.5345
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Low Back Pain; Mechanical Low Back Pain; Backache
Keywords: Low back pain; Thrust manipulation; Spinal manipulation; Joint mobilization; Non-thrust manipulation; proprioception; Postural stability; Baropodometry
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Manipulation, Spinal; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrust manipulation (TM) (Experimental): The patients allocated to the TM group will receive TM aimed at the L4-L5 intervertebral segments. All the patients will be positioned in a standardized position (right side-lying) and will receive a rotational TM technique. The treating therapist will have up to two attempts to perform the TM in each patient.
  There is no need for cavitation in order to consider the TM successful; the occurence of cavitation, however, will be recorded.
  A single treatment will be provided.
  Interventions: Other: Thrust Manipulation
- Non-thrust manipulation (NTM) (Experimental): The patients allocated to the NTM group will receive TM aimed at the L4-L5 intervertebral segments. All the patients will be positioned in a standardized position (right side-lying) and will receive 30 oscilations of a grade III rotational NTM.
  A single treatment will be provided
  Interventions: Other: Non-thrust manipulation (NTM)

INTERVENTIONS:
Other: Thrust Manipulation — After positioning patients in right side-lying, a rotational TM technique will be addressed at the L4-L5 lumbar segments. The treating therapist will have up to two attempts to apply the TM.
  Other Names: Spinal manipulation; Lumbar manipulation; Lumbar thrust; Manual Therapy; Manipulative therapy
  Arms: Thrust manipulation (TM)
Other: Non-thrust manipulation (NTM) — A grade III rotational non-thrust manipulation will be addressed at the L4-L5 lumbar segments. Thirty oscilations will be performed.
  Other Names: Mobilization; Joint mobilization; lumbar mobilization; Manual therapy; Maitland
  Arms: Non-thrust manipulation (NTM)

SUMMARY:
This study aims to verify the effects of Thrust Versus Non-thrust Manipulation on Pain, Trunk Proprioception and Postural Stability in Subjects With Chronic Low Back Pain.

DETAILED DESCRIPTION:
Forty individuals with chronic low back pain will be randomly assigned, by a researcher not involved in data collection, to two treatment groups: Thrust manipulation (side-lying rotational manipulation standardized to the L4-L5 level) or non-thrust manipulation (side-lying grade III rotational non-thrust manipulation). A single treatment session will be provided.

Outcome measurement will be conducted immediately after the treatment session. Data will be collected by a blinded assessor. Between-group differences will be calculated by constructing mixed linear models following an intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Chronic Low back pain (pain lasting for at least 12 weeks)
* NPRS ≥ 3

Exclusion Criteria:

* Previous surgery or fracture at the lumbar spine
* Pregnancy
* Inflammatory disorders
* Symptoms distal to the gluteal line
* Having received manipulative treatment in the past four weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain | Up to 10 minutes after intervention
  Pain will me measured Up to 10 minutes after intervention by an 11 point (0-11) Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Global Perceived Effect | Up to 10 minutes after intervention
  Global Perceived effect will be measured by an 11 point (-5-+5) Global Perceived Effect (GPE)
Lumbar joint position sense | Up to 10 minutes after intervention
  Lumbar joint position sense will be measured by a isokinetic dynamometer (BIODEX System 4 Pro™, Shirley, NY)
Peak plantar pressure | Up to 10 minutes after intervention
  Peak plantar pressure will be measured by a digital baropodometer (FootWork Pro)
Center of Pressure displacement | Up to 10 minutes after intervention
  CoP displacement will be measured by a digital baropodometer (FootWork Pro) by means of stabilometry

OTHER OUTCOMES:
Foot contact area | Up to 10 minutes after intervention
  Foot contact area will be measured by a digital baropodometer (FootWork Pro)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Silva, PhD, Study Chair — Adjunct professor
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil